CLINICAL TRIAL: NCT01351571
Title: An Open Label, Prospective, Observational, Non-interventional Study of Bevacizumab in Combination With Interferon Alpha-2a for the First-line Treatment of Patients With Advanced and/or Metastatic Renal Cell Carcinoma
Brief Title: An Observational Study of Avastin (Bevacizumab) in Combination With Interferon Alpha-2a as First-Line Treatment in Patients With Advanced and/or Metastatic Renal Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25251
Record Dates: First submitted 2011-05-09; First posted 2011-05-11 (Estimated); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational study will evaluate the safety and efficacy of Avastin (bevacizumab) in combination with interferon alpha-2a as first-line treatment in patients with advanced and/or metastatic renal cell carcinoma. Data will be collected from each patient as per routine clinical practice of the Investigator (maximum of 52 weeks, until disease progression /unacceptable toxicity or withdrawal of consent) and/or based on the local label.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Advanced and/or metastatic renal cell carcinoma
* Receiving first-line treatment with Avastin and interferon alpha-2a according to standard of care and current local label
* At least one measurable and non-measurable lesion according to RECIST criteria
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Adequate bone marrow, renal and liver function

Exclusion Criteria:

* Contraindications to Avastin and/or interferon alpha-2a as per local label

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced and/or metastatic renal cell carcinoma treated with Avastin and interferon alpha-2a
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2010-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | approximately 4 years

SECONDARY OUTCOMES:
Progression-free survival: time from first drug administration to documented disease progression or death of any cause | approximately 4 years
Overall response rate: complete response or partial response according to RECIST criteria | approximately 4 years
Overall survival | approximately 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- India (2):
  - Aurangabad
  - Delhi